CLINICAL TRIAL: NCT04978077
Title: Networks of Bacterium-Metabolite Interactions in the Small Intestine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of the specific study population consisting of stoma patients proved escpecially difficult, so the recruitment was halted before the anticipated target number
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-01108
Record Dates: First submitted 2021-07-12; First posted 2021-07-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diet, Healthy; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat test meal first, high carbohydrate test meal second (Experimental): Consumption of a high fat challenge first, consumption of a high carbohydrate challenge after two weeks wash out
  Interventions: Other: Test meal (high fat = Nutricia Calogen®, or high carbohydrate = Nutricia preOp®)
- High carbohydrate test meal first, high fat test meal second (Experimental): Consumption of a high carbohydrate challenge first, consumption of a high fit challenge after two weeks wash out
  Interventions: Other: Test meal (high fat = Nutricia Calogen®, or high carbohydrate = Nutricia preOp®)

INTERVENTIONS:
Other: Test meal (high fat = Nutricia Calogen®, or high carbohydrate = Nutricia preOp®) — After a night fast participants will drink the test meal

SUMMARY:
Probands with an Ileo- or Colostomy are assigned to consume a test meal which is either high in fat or high in carbohydrates. After the test meal samples from the stoma, urine, blood and skin are retrieved. These will be subjected to large scale analyses of microbiota and metabolite content. To get a better comparability test subjects will consume a standardized liquid diet three days before the study day.

DETAILED DESCRIPTION:
Between both study days a two week wash out phase will be done. During the study day sampling will be done at set time points until 8 hours after the consumption of the test meal.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* General good health
* Ileostomy or colostomy

Exclusion Criteria:

* Hematologic disorders with contraindication of blood draw
* Participation in other clinical trial interfering with study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Identification of stimulating and inhibiting metabolite and bacteria interactions | 8 hours
  Correlation of results of secondary outcome measures to find interactions
Reproduction of metabolite-bacteria interactions in vitro culture | 2 weeks
  By culturing of bacteria with possible interactions together in vitro

SECONDARY OUTCOMES:
Analysis of bacteria species composition | 8 hours
  by 16S rRNA sequencing of sample content
Cultivation of bacterial strains in various conditions including ileal fluids | 2 weeks
  Cultivation of native species found in samples, as well as dedicated E. coli with recording capacity for transcriptional changes
Metabolite composition in intestinal fluids | 8 hours
  by untargeted mass spectrometry
Metabolite composition in blood | 8 hours
  by untargeted mass spectrometry
Metabolite composition in urine | 8 hours
  by untargeted mass spectrometry
Metabolite composition in intestinal fluids, blood and urine | 8 hours
  by untargeted mass spectrometry
Analyze eucaryotic and viral microbiome composition | 8 hours
  by shotgun sequencing of sample content
Analysis of microbiota metabolic potential | 8 hours
  by shotgun sequencing of sample content
Analysis of microbiota metabolic activity | 8 hours
  by sequencing of transcriptome of sample content
Analysis of microbiota biomass | 8 hours
  by measuring absolute bacteria counts by flow cytometry of 16S spiking

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, Prof. Dr. med., Principal Investigator — University Clinic for Visceral Surgery and Medicine
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be shared in a public repository
Time Frame: upon publication of study results open ended
Access Criteria: public access